CLINICAL TRIAL: NCT03269656
Title: Association of Pre-diagnostic Vitamin D Levels and Survival in Older Individuals With Cancer
Brief Title: Age Gene/Environment Susceptibility Reykjavik Study
Acronym: AGES
Status: Completed | Type: Observational
Sponsor: Icelandic Heart Association (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Sponsor
Other Study IDs: IHA; NO1-AG-1-2100 (Other Grant/Funding Number: National Institute on Aging); ZIAEY000401 (NIH)
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Neoplasms
Keywords: Vitamin D; Cancer; Survival
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AGES-Reykjavik participants: Exploring whether pre-diagnostic serum levels of 25(OH)D among older individuals living in Iceland were associated with survival after cancer diagnosis. We also assessed the risk of being diagnosed with cancer in association with 25(OH)D levels.

SUMMARY:
5764 men and women in Iceland, aged 66 to 96 years entered the Ages Gene/Environment Susceptibility (AGES) - Reykjavik Study. Serum 25(OH)D was measured in 5,519 of all 5,764 (96%) participants at study entry in year 2002 through 2006. The main emphasis was on exploring whether pre-diagnostic serum levels of 25(OH)D were associated with survival after cancer diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* To participate in the AGES-Reykjavik study

Exclusion Criteria:

* To be diagnosed with cancer before study entry

Ages: 66 Years to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In 1967, all 30,795 men and women living in the capital area of Iceland and born between 1907 and 1935 were invited by the Icelandic Heart Association to join a prospective cohort study. Approximately 19,000 attended the clinic at least once and became participants of the Reykjavik Study. Subsequently, in 2002, a random sample of the cohort comprising 5,764 men and women who were still alive in Iceland and aged 66 to 96 years entered the Ages Gene/Environment Susceptibility (AGES) - Reykjavik Study
Sampling Method: Probability Sample
Enrollment: 5764 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2006-01-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of diagnosis until death or censored at end of the follow-up (December 31, 2014)
  The association between pre-diagnostic 25(OH)D levels in cancer patients and overall survival
Cancer survival | From date of diagnosis until cancer death or censored at the end of the follow-up (December 31, 2014)
  The association between pre-diagnostic 25(OH)D levels in cancer patients and cancer survival

SECONDARY OUTCOMES:
Cancer diagnosis | From date of blood draw (study entry) until cancer diagnosis, death or end of the observation period (December 31, 2014) whichever occurred first
  The association between pre-diagnostic 25(OH)D levels and cancer risk

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Torfadottir, PhD, Principal Investigator — University of Iceland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harris TB, Launer LJ, Eiriksdottir G, Kjartansson O, Jonsson PV, Sigurdsson G, Thorgeirsson G, Aspelund T, Garcia ME, Cotch MF, Hoffman HJ, Gudnason V. Age, Gene/Environment Susceptibility-Reykjavik Study: multidisciplinary applied phenomics. Am J Epidemiol. 2007 May 1;165(9):1076-87. doi: 10.1093/aje/kwk115. Epub 2007 Mar 10. PMID 17351290
- See also: Age, Gene/Environment Susceptibility-Reykjavik Study: Multidisciplinary Applied Phenomics — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2723948/